CLINICAL TRIAL: NCT05750940
Title: Oxidative Skeletal Muscle Metabolism in Chronic Heart Failure Patients With and Without Iron Deficiency
Acronym: FERRIFY
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Peter van der Meer, MD PhD, Prof. dr. Peter van der Meer, University Medical Center Groningen
Other Study IDs: 201700917
Record Dates: First submitted 2021-10-05; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: HF - Heart Failure; Iron-deficiency
Keywords: 31P MRS; 31Phosphor Magnetic Resonance Spectroscopy; HFpEF; HFrEF; Oxidative Skeletal Muscle Metabolism
MeSH Terms: conditions — Heart Failure; Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 31Phosphor Magnetic Resonance Spectroscopy — Measurement of skeletal oxidative metabolism with 31phosphor magnetic resonance spectroscopy

SUMMARY:
Observational study using in vivo noninvasive 31 phosphor magnetic resonance spectroscopy (31P MRS) to quantify the effect of iron deficiency (ID) on skeletal oxidative metabolism in patients with chronic heart failure (HF).

DETAILED DESCRIPTION:
Iron Deficiency (ID) is a comorbidity in heart failure (HF) patients with high prevalence and severe clinical consequences. Multiple studies have shown that ID in HF patients impairs exercise capacity, quality of life and outcome. It is currently unknown whether these detrimental consequences of ID are due to cardiovascular or hematologic effects, or deteriorated peripheral muscle metabolism and function. This study was designed to quantify the effect of ID on skeletal oxidative metabolism in patients with chronic HF.

ELIGIBILITY:
Inclusion Criteria:

For HFrEF patients:

* Diagnosis of chronic HF of either ischemic or non-ischemic etiology;
* Stable, evidence-based medical therapy for HF;
* LVEF <40% measured <5 year prior to inclusion;
* NYHA class II - III (symptomatic HF) at moment of inclusion;

For HFpEF patients:

* Diagnosis of chronic HF of either ischemic or non-ischemic etiology;
* LVEF >40% and one of the following parameters, measured <5 year prior to inclusion;
* Left atrial volume index (LAVI) >34 mL/m2 or
* left ventricular mass index ≥115 g/m2 (for males) or ≥95 g/m2 (for females) or
* E/e' ≥13 or
* mean e' (septal and lateral) <9 cm/s
* NYHA class II - III (symptomatic HF) at moment of inclusion;
* Serum NT-proBNP ≥125 pg/mL when in sinus rhythm; >300 pg/mL when in atrial fibrillation.

Additional inclusion criterion for subjects with ID:

- Iron deficiency, defined as TSAT <20%.

Exclusion Criteria:

* Age <18 years;
* Unable or unwilling to undergo exercise MRI (e.g. pregnancy, physical disabilities, claustrophobia);
* The presence of ferromagnetic material in/on the body which cannot be removed (e.g. non-MRI-compatible cardiac devices, tattoos containing ferrous ink);
* History of erythropoietin stimulating agent, intravenous iron therapy and/or blood transfusion <3 months prior to study enrolment;
* Moderate anaemia, defined as Hb <7 mmol/L for both men and women;
* Oral iron therapy >100 mg/day <4 weeks prior to study enrolment;
* Unable to understand study procedures;
* Unable or unwilling to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For this study, we will include 40 non-anaemic patients with stable chronic HF, subdivided in 20 patients with HFrEF and 20 subjects with HFrEF. HFpEF and HFrEF patients will be further subdivided into 10 patients with ID and 10 patients without ID. These patients will be recruited from the outpatient clinic of the Department of Cardiology, UMCG. Patients must be stable at the time of inclusion (i.e. no medication changes <1 month prior to study).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-10-05 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
ΔPi/PCr from baseline to maximum exercise | During study visit, from resting baseline to maximum exercise (from start exercise upto exhaustion for a maximum timeframe of 10 minutes)
  Δ ratio of inorganic phosphate/Phosphocreatinin concentrations from baseline to maximum exercise

SECONDARY OUTCOMES:
PCr recovery rate during recovery | During study visit, from maximum exercise to end of recovery (upto at least 5 minutes after end of exercise)
  Post-exercise phosphocreatinin recovery rate
Intramuscular pH | During study visit, during exercise (from start exercise upto exhaustion for a maximum timeframe of 10 minutes)
  Rates and magnitude of change in intramuscular pH during exercise
Maximal exercise performance | During study visit, during exercise (from start exercise upto exhaustion for a maximum timeframe of 10 minutes)
  Maximal exercise performance

CONTACTS AND LOCATIONS:
Locations (1):
- UMCG, Groningen, Netherlands